CLINICAL TRIAL: NCT06646302
Title: Neural and Clinical Effects of 40 Hz Burst Stimulation in Tinnitus: a Four-phase Self-controlled Study
Brief Title: Residual Inhibition of 40 Hz Burst Sound in Tinnitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024087
Record Dates: First submitted 2024-10-09; First posted 2024-10-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus
Keywords: Tinnitus; 40 Hz stimulation; Acoustic therapy; Residual inhibition; Personalized medicine
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Personalized 40 Hz Broadband Stimulation (Experimental): Participants receive personalized broadband acoustic stimulation modulated at 40 Hz. An adaptive equalization algorithm, based on individual and population residual inhibition (RI) responses, is used to weight frequency components across 125 Hz-12 kHz.
  Interventions: Other: Personalized 40 Hz Broadband Stimulation
- 40 Hz Pure Tone Stimulation (Experimental): Participants receive pure tone stimulation at the individually optimized carrier frequency identified in earlier phases, amplitude-modulated at 40 Hz.
  Interventions: Other: 40 Hz Pure Tone Stimulation
- Continuous Broadband Noise (Active Comparator): Participants receive continuous broadband noise stimulation without 40 Hz modulation.
  Interventions: Other: Continuous Broadband Noise

INTERVENTIONS:
Other: Personalized 40 Hz Broadband Stimulation — Broadband acoustic stimulus (125 Hz-12 kHz) amplitude-modulated at 40 Hz with a 50% duty cycle. A polynomial regression and FFT-based algorithm applies individualized frequency weighting, combining population data (70%) and patient-specific responses (30%). Delivered for 60 seconds at 10 dB above the individual minimum masking level (MML).
  Arms: Personalized 40 Hz Broadband Stimulation
Other: 40 Hz Pure Tone Stimulation — Pure tone stimulus at the optimized frequency (matched to tinnitus characteristics or high-frequency carrier), amplitude-modulated at 40 Hz with a 50% duty cycle. Delivered for 60 seconds at 10 dB above MML.
  Arms: 40 Hz Pure Tone Stimulation
Other: Continuous Broadband Noise — Continuous broadband noise spanning 125 Hz-12 kHz without 40 Hz modulation. Delivered for 60 seconds at 10 dB above MML as an active control condition.
  Arms: Continuous Broadband Noise

SUMMARY:
Tinnitus affects 10-15% of adults and is frequently associated with impaired quality of life, anxiety, and sleep disturbance. Conventional sound therapies based on continuous masking provide inconsistent and short-lived relief, and the neural mechanisms underlying residual inhibition (RI) remain unclear.

This study aims to determine whether 40 Hz burst stimulation with high-frequency carriers can achieve longer-lasting RI than continuous sound, and to explore its underlying neural mechanisms using EEG.

DETAILED DESCRIPTION:
Residual inhibition (RI) refers to the temporary reduction or disappearance of tinnitus following sound stimulation and provides an important clue for identifying patients who may benefit from acoustic therapy. However, the effects of different sound stimulation strategies on RI remain poorly understood.

This study evaluates whether 40 Hz burst-modulated sound achieves stronger and longer RI compared with conventional continuous stimulation. The trial follows a four-phase design:

Phase 1: Exploratory testing of burst versus continuous tones at different frequencies.

Phase 2: Large-scale validation in 265 patients. Phase 3: Development of a personalized stimulation protocol using adaptive spectral optimization.

Phase 4: EEG investigation of neural mechanisms, focusing on gamma oscillations and functional connectivity changes.

The primary outcomes are the strength and duration of tinnitus suppression. Secondary outcomes include EEG markers such as γ-band power spectral density and phase-locking value.

By combining behavioral and neurophysiological measures, this study aims to establish 40 Hz burst stimulation as a novel rhythm-based sound therapy and to provide mechanistic insights that may enable more effective, personalized tinnitus management.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with subjective tinnitus;
2. Chronic tinnitus: tinnitus course ≥ 1 month;
3. Normal middle ear function;
4. The average hearing threshold (defined as mean of 0.5, 1, 2, and 4 kHz) of the unaffected ear < 60 dB;
5. Tinnitus can be heard under normal circumstances.
6. Subjects are able to understand the purpose of the study, volunteer to participate and cooperate with the instructors to complete the experiment, and be willing to sign the informed consent.

Exclusion Criteria:

1. Acute phase tinnitus;
2. Fluctuating tinnitus loudness;
3. Severe psychiatric disorders;
4. Inability to complete tinnitus testing;
5. Fluctuating or retrocochlear hearing loss;
6. Conductive hearing loss;
7. Currently participating in other research projects that may affect tinnitus;
8. Subjects who are not considered suitable for this clinical trial by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Tinnitus suppression strength | Immediately after the sound stimulation session.
  Residual inhibition depth, 0-100% reduction
Residual inhibition duration | Immediately after the sound stimulation session.
  Time in seconds until tinnitus returns to baseline after stimulation

SECONDARY OUTCOMES:
EEG spectral power changes | measured across the entire 10-minute EEG recording session (baseline, during stimulation, and post-stimulation)
EEG functional connectivity changes | measured across the entire 10-minute EEG recording session (baseline, during stimulation, and post-stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, PhD, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No